CLINICAL TRIAL: NCT05226130
Title: Non-invasive Vagal Nerve Stimulation to Improve Functional Outcomes in Veterans With Alcohol Use Disorder
Brief Title: Non-invasive Vagal Nerve Stimulation in Alcohol Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3629-M
Record Dates: First submitted 2021-12-27; First posted 2022-02-07 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use; neuromodulation; neuroimaging; withdrawal; anxiety; quality of life
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Devices include a sham and an active noninvasive vagal nerve stimulator (nVNS). Devices are identical in appearance, and both produce reliable sensation on the skin when applied to the neck area (transcutaneous cervical stimulation). Stimulation duration is approximately 120 seconds for both sham and active devices. Subjects receive the same instructions to self-administer stimulation twice a day for 120 minutes on each side (right and left).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the research team involved in data collection and subjects will be blinded (double-blind study design). Subjects will be randomly assigned to receive either active or sham stimulation. Devices will be marked with an identification number to mask treatment condition. An unblinded Co-Investigator, not involved in data collection and subject contact, will assign randomization, provide device identification number, and keep the key linking condition to identification numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active cervical transcutaneous vagus nerve stimulation (Active Comparator): Participants will be assigned to active transcutaneous vagus nerve stimulation, received once during each of the study visits and self-administered twice a day for a week.
  Interventions: Device: Cervical transcutaneous vagus nerve stimulation (active comparator)
- Sham cervical transcutaneous vagus nerve stimulation (Placebo Comparator): Participants will be assigned to sham transcutaneous vagus nerve stimulation, received once during each of the study visits and self-administered twice a day for a week.
  Interventions: Device: Cervical transcutaneous vagus nerve stimulation (sham comparator)

INTERVENTIONS:
Device: Cervical transcutaneous vagus nerve stimulation (active comparator) — Active nVNS produces low-voltage electrical signal that generates sensations on the skin on upper anterior cervical area (overlying carotid artery) and that stimulates the vagus nerve.
  Arms: Active cervical transcutaneous vagus nerve stimulation
Device: Cervical transcutaneous vagus nerve stimulation (sham comparator) — Sham nVNS produces low-voltage electrical signal that generates sensations on the skin on upper anterior cervical area (overlying carotid artery) and that does not stimulate the vagus nerve.
  Arms: Sham cervical transcutaneous vagus nerve stimulation

SUMMARY:
Alcohol use disorder (AUD) is a major health concern amongst Veterans as it causes poor health, lost days at work, impaired psychosocial functioning, and decreased quality of life. Current treatment options for AUD show limited effectiveness, which is exemplified by high relapse rates. Chronic heavy drinking results in psychological and physical distress during abstinence, including anxiety, irritability, and general discomfort, which increases the urge to drink to relieve these symptoms. The hypothesis of this study is that noninvasive vagal nerve stimulation (nVNS) can modify the perception of such inner bodily sensations of distress, and consequently reduces the drive to drink for relief. The aim of this study is to establish feasibility and acceptability of applying nVNS as a rehabilitative treatment for AUD in Veterans. The study will also evaluate the effect of nVNS on functional outcomes, quality of life, distress, and craving, and if nVNS alters neural activation patterns in brain regions involved in the perception and awareness of distress and pain.

DETAILED DESCRIPTION:
AUD is a serious mental health disorder that affects more than 40% of US military Veterans, presenting a major burden to this population. Relapse rates of AUD are extremely high; over half of Veterans who complete treatment, relapse within 6 months, highlighting the need for improved treatments or differing treatment targets. Chronic, heavy drinking leads to an imbalance in homeostasis resulting in psychological and physical distress during periods of abstinence, and the urge to drink to relieve these symptoms to restore homeostasis.

nVNS is a low-risk form of neuromodulation that has been shown to alleviate anxiety and chronic pain, and to reduce drug and alcohol relapse in animal models. The investigators hypothesize that nVNS attenuates distress-related craving in AUD in humans by modifying the autonomic nervous system and changing the perception of inner bodily sensations of physiological and affective distress. The investigators also hypothesize that nVNS improves functional outcomes and quality of life in Veterans with AUD.

The proposed research will include 16 Veterans who meet for a diagnosis of AUD. Subjects will be randomly assigned to receive nVNS or sham stimulation prior to performing a well-validated functional Magnetic Resonance Imaging task designed to assess neural correlates of physical distress (via a heat stimulus). Subjects will then self-administer nVNS/sham at home twice a day for 7 days and return for a follow-up visit, during which all study components will be repeated. Behavioral assessments of functional disability, quality of life, psychological and physiological distress, and craving will be administered at baseline, after stimulation, and at follow-up.

The aim of the proposed study is to establish feasibility and acceptability of applying nVNS as a rehabilitative treatment for AUD. In addition, the study will evaluate the preliminary effectiveness of nVNS in improving functional outcomes and quality of life, in reducing distress and craving, and in altering neural activation patterns in brain regions involved in the perception and awareness of distress and pain. The proposed work has the potential to lead to innovative, low-risk treatment options with high promise to significantly improve the care and lives of Veterans as there is a need for alternative treatments for AUD. As such, this novel AUD treatment could be particularly beneficial for Veterans who do not tolerate pharmacotherapy, and who have access or cognitive limitations or stigma concerns that act as barriers to psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Male subjects between 21 and 65 years of age
* Current DSM-5 diagnosis of AUD with at least one functional disability due to alcohol use, current alcohol craving, and current heavy drinking (>4 drinks on any day or >14 drinks per week)
* Able to forgo consumption of alcohol for 24 hours without any serious discomfort including nausea/vomiting, visual/auditory/tactile hallucinations, or non-essential tremor

Exclusion Criteria:

* Clinical Institute Withdrawal Assessment of Alcohol Scale (CiWA) score >=9 on the day of the scan (symptoms judged to be due to co-existing anxiety or headache disorders will not be counted toward the total).
* Currently or recently (within last 90 days) enrolled in abstinence-based treatment program.
* Evidence of a maladaptive pattern of substance use or abuse other than alcohol one month prior to screening visit.
* Severe mental illness, e.g., psychosis or bipolar disorder
* At risk for suicide or homicide
* History of neurological disorder that might be associated with cognitive dysfunction.
* History of head trauma involving loss of consciousness >24 hours
* Clinically significant uncontrolled/unstable medical illness or clinically significant surgery within 1 month of the screening visit.
* MRI-related exclusion criteria: cardiac pacemaker, metal fragments in eyes/skin/body, aortic/aneurysm clips, heart-valve replacement, copper intrauterine device, shunt (ventricular or spinal), neuro/bio-stimulators
* Vagus nerve stimulation related criteria: history of carotid endarterectomy, severe carotid artery disease (e.g., history of transient ischemic attack (TIA) or stroke], congestive heart failure, cardiac arrhythmia, known severe coronary artery disease or recent myocardial infarction (within 5 years), history of seizure or syncope (within past year), prior neck surgery.

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Parent study does not enroll women (due to potential sex differences in inflammation-induced alterations of brain response as well as sex differences in prevalence of PTSD), this study will not enroll women either to allow for post-hoc group comparisons. If significant effects are demonstrated with this study, follow-up grant proposals will include females.
Enrollment: 19 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Klaming, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Started | 9 | 10
Completed | 9 | 7
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Not treatment adherent | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (8.6) | 39.6 (7.2) | 38.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 1 | 3
  White | 6 | 4 | 10
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Treatment Acceptability Questionnaire (TAQ)
Description: The Treatment Acceptability Questionnaire (TAQ) is a self-rating questionnaire used to assess acceptability of a treatment. The TAQ uses a 7-point rating scale ranging from 1 to 7, with lower scores reflecting lower acceptability and a midpoint of 4 indicating neutral acceptability. A rating above the midpoint of the TAQ (i.e., score between 5 and 7) is the established criterion for "acceptable to highly acceptable".
Time Frame: Measure administered at study completion (i.e., 1 week after baseline)
Population: TAQ ratings for two subjects (both in the sham group) were not included in the analyses because they were not treatment adherent (i.e., did not self-administer nVNS/sham as instructed). One subject was lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 7
score on a scale | 5.7 (1.0) | 6.4 (0.8)

2. Primary Outcome: Measurement of Feasibility - Recruitment Goal (Data Reflects the Number of Participants Who Were Successfully Enrolled in the Study)
Description: Treatment feasibility will be evaluated by meeting the proposed recruitment goal of 16 Veterans within 12 months. This aim was measured as the number of study participants who signed the study consent form, completed at least the baseline study visit, and were included in the study analyses.
Time Frame: Baseline
Population: More (19 subjects) than the initially proposed number of participants (16 subjects) were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 10
Participants | 9 | 10

3. Primary Outcome: Measurement of Feasibility - Treatment Adherence (Number of Times Subjects Self-administered nVNS/Sham Stimulation for 7 Days as Instructed)
Description: Treatment adherence will be assessed via a daily treatment completion log, and calculated by dividing the total number of times subjects were instructed to self-administer the nVNS/sham stimulation (2x/day for 7 days = 14 times) by the number of times the subjects actually self-administered the stimulation. Treatment feasibility will be evaluated by meeting >75% treatment adherence during the 1-week interval.
Time Frame: Baseline to week 1 of 2x daily intervention
Population: 1 subject lost to FU
Measure: Mean (Standard Deviation); unit: percentage of treatment administrations
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 9
percentage of treatment administrations | 94.4 (7.8) | 79.76 (26.4)

4. Primary Outcome: Measurement of Feasibility - Subject Retention (Number/Percentage of Subjects Who Return for a Follow-up Visit)
Description: Treatment feasibility will be evaluated by meeting >75% subject retention at follow-up as measured by the number/percentage of subjects who return for a follow-up visit and complete primary outcome measures and return the device to the study team.
Time Frame: Baseline to post treatment, up to 21 days post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 10
Participants | 9 | 9

5. Primary Outcome: Measurement of Feasibility - Serious Adverse Side Effects
Description: Treatment feasibility will be evaluated by no occurrence of serious adverse side effects (as documented in checklist/daily log, interview at study completion, or otherwise reported by the participant).
Time Frame: Baseline to week 1 of 2x daily intervention
Population: Number of serious adverse events
Measure: Number; unit: Number of serious adverse events
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 10
Number of serious adverse events | 0 | 0

6. Secondary Outcome: Substance Use Recovery Evaluator (SURE)
Description: The Substance Use Recovery Evaluator (SURE) assesses the following domains of AUD-related functional outcomes: self-care (mental and physical health), relationships, material resources (stability of housing and occupational resources), and outlook of life. The SURE has been developed for use in substance use disorder populations. The SURE is comprised of 21 items, rated on a 3-point scale, but scored using a 3-point scale. Scores range from 21-63. A higher score indicates better functional outcomes.
Time Frame: Baseline to week 1 of 2x daily intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 44.7 (7.8) | 44.0 (5.7)
  Follow-up | 50.6 (10.5) | 44.9 (8.8)

7. Secondary Outcome: WHO Quality of Life Assessment (WHOQOL-BREF) - Psychological Domain
Description: The WHO Quality of Life assessment (WHOQOL-BREF) assesses quality of life across four domains (physical health, psychological, social relationships, and environment) with a total of 26 questions. The rating scale ranges from 1 to 5 and minimum and maximum values varies between domains (physical health: 7-35, psychological: 6-30, social relationships: 3-15, environment: 8-40). Higher scores denote higher quality of life. Reported here are results from the psychological domain.
Time Frame: Baseline to week 1 of 2x daily intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 14.2 (4.1) | 17.8 (4.0)
  Follow-up | 16.8 (4.4) | 17.4 (4.3)

8. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The Beck Anxiety Inventory (BAI) is a self-report instrument to measure the severity of anxiety and emotional distress. The BAI is a 21-item questionnaire with a 4-point rating scale (0-3), with a higher score reflecting greater anxiety. Total scores range from 0 to 63 with higher scores indicating higher anxiety.
Time Frame: Baseline to week 1 of 2x daily intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 16.8 (9.2) | 17.0 (11.6)
  Follow-up | 12.5 (10.0) | 17.6 (17.8)

9. Secondary Outcome: PROMIS Pain Interference
Description: The PROMIS Pain Interference measures self-reported consequences of pain on relevant aspects of one's life, i.e., the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. This questionnaire has 8 items with ratings ranging from "not at all" to "very much". Total score minimum is 8 and the maximum is 40. Higher scores reflect higher interference of pain with level of functioning.
Time Frame: Baseline to week 1 of 2x daily intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 22.4 (8.3) | 23.6 (9.7)
  Follow-up | 20.9 (8.2) | 21.8 (11.0)

10. Secondary Outcome: Alcohol Urge Questionnaire (AUQ)
Description: The Alcohol Urge Questionnaire (AUQ) is 8-item scale that measures cognitive preoccupation with alcohol on a 7-point rating scale ranging from "strongly disagree" to "strongly agree". Two items are reverse scored. Minimum score is 8 and maximum is 56. Higher scores reflect greater craving.
Time Frame: Baseline to week 1 of 2x daily intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 25.6 (11.3) | 25.7 (10.8)
  Follow-up | 18.4 (9.8) | 21.2 (8.3)

11. Other Pre Specified Outcome: Neural Response to Heat Pain Stimuli (Measured as Sum of BOLD Beta Coefficients Over Time in Arbitrary Units)
Description: Participants receive brief thermal stimuli (experienced temperature ranging from warm to hot) applied to the leg via a contact thermode during a functional magnetic resonance imaging scan. Neural activation will be measured using the general linear model (GLM) to estimate beta coefficients for the BOLD (blood-oxygen-level-dependent) signal in response to thermal stimulation. Activation in the brain region insula will be summarized by calculating the area under the beta response curve (arbitrary units) over the stimulus duration (i.e., time), reflecting the total magnitude of neural activation. BOLD signal and beta coefficients used to model neural response are in arbitrary units. The area under the curve is the cumulative scaled beta (i.e., cumulative percent signal change) that is most reflective of the activation attributable to the stimulus. Higher numbers indicate more neural activation in the insula in response to painful heat stimuli.
Time Frame: Baseline to week 1 of 2x daily intervention
Population: Two subjects did not participate in neuroimaging scans due to claustrophobia.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
Number analyzed (Participants) | 9 | 8
Arbitrary units
  Baseline | -0.48 (0.25) | -0.37 (0.27)
  Follow-up | -0.38 (0.24) | 1.00 (1.21)

ADVERSE EVENTS:
Time Frame: 7 days
Description: [Not Specified]
Arm/Group | Active Cervical Transcutaneous Vagus Nerve Stimulation | Sham Cervical Transcutaneous Vagus Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 4/9 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Cervical Transcutaneous Vagus Nerve Stimulation (N=9) | Sham Cervical Transcutaneous Vagus Nerve Stimulation (N=10)
Lip pulling (Product Issues) | 2 (2) | 0 (0)
Tingling sensation (Product Issues) | 2 (2) | 0 (0)
Muscle twitching (Product Issues) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mild headache (Nervous system disorders) | 1 (1) | 0 (0)
Neck soreness (Product Issues) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT05226130/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT05226130/ICF_000.pdf